CLINICAL TRIAL: NCT01239368
Title: Rapamycin-Resistant T Cell Therapy of Multiple Myeloma: Relapse Prevention and Relapse Therapy
Brief Title: Th1/Tc1 Immunotherapy Following Stem Cell Transplantation in Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Hackensack Meridian Health (Other); Georgetown University (Other)
Responsible Party: Principal Investigator, Steven Pavletic, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110016; 11-C-0016
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Myeloma, Plasma-Cell; Myeloma-Multiple; Myelomatosis
Keywords: Multiple Myeloma; High Risk; Newly Diagnosed; Adoptive Immunotherapy; Autologous
MeSH Terms: conditions — Multiple Myeloma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort B - Relapsed Multiple Myeloma (Experimental): Th1 (type 1 T helper cells)/Tc1 (T cytotoxic cells, type 1) .Rapamycin (Rapa) for Relapsed Multiple Myeloma
  Interventions: Procedure: Adoptive Immunotherapy; Biological: Th1/Tc1 Rapa Cell Therapy
- Cohort A - Prevention of Relapse (Experimental): Th1/Tc1.Rapa Prevention of Relapse
  Interventions: Procedure: Adoptive Immunotherapy; Biological: Rapamycin-Generated Autologous Th1/Tc1 Cells (modified primary human T cells); Biological: Th1/Tc1 Rapa Cell Therapy

INTERVENTIONS:
Procedure: Adoptive Immunotherapy — Th1 (type 1 T helper cells)/Tc1 (T cytotoxic cells, type 1) Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
Biological: Rapamycin-Generated Autologous Th1/Tc1 Cells (modified primary human T cells) — Six Th1/Tc1 Rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Arms: Cohort A - Prevention of Relapse
Biological: Th1/Tc1 Rapa Cell Therapy — Th1/Tc1Rapa: 5 x 10e(6) cells/kg

SUMMARY:
Background:

- Cancer development is associated with problems in immune system functions, which prevent the body from attacking and destroying the abnormal cells that lead to tumor growth. Research has suggested that certain white blood cells, known as Th1 (type 1 T helper cells) and Th2 T cells (type 2 T helper cells), are affected in individuals with some kinds of cancer -- when the proportion of Th2 cells is greater than Th1 cells, the immune systems ability to fight off the growth of malignant tumors is weakened. Researchers are interested in determining if an infusion of specially modified Th1 cells, in addition to stem cell transplant, is a safe and effective treatment for individuals with forms of multiple myeloma that might not respond well to standard treatments alone.

Objectives:

- To determine the safety and effectiveness of the infusion of modified Th1 white blood cells, in conjunction with standard treatment, as a treatment for individuals who have been diagnosed with high-risk forms of multiple myeloma.

Eligibility:

* Individuals age 18 to 75 who have been newly diagnosed with high-risk multiple myeloma and who have received no or minimal treatment (Cohort A).
* Individuals age 18 to 75 who have relapsed multiple myeloma, as defined by measurable disease after at least 2 prior treatment regimens.

Design:

* Participants will be screened with a medical history, physical examination, blood and urine tests, and imaging studies. Some participants may also have a bone marrow or other type biopsy to evaluate the state of their disease.
* White blood cells will be collected from the participants through an apheresis procedure, which will collect and separate the white blood cells and return the rest of the blood to the participant.
* The collected cells will be grown and expanded under special conditions in the laboratory and stored frozen until participants receive standard of care treatment for multiple myeloma, including a stem cell transplant.
* Participants will receive an infusion of the modified Th1 cells a few weeks after the transplant, and will remain in the hospital for a few days after receiving the cells to monitor the possible immediate effects of the treatment.
* Participants will have regular follow-up visits to study the long-term effects of the modified Th1 cell infusion.

DETAILED DESCRIPTION:
Background:

* Autologous Hematopoietic Cell Transplantation (AHCT), which represents the standard of care for newly diagnosed Multiple Myeloma (MM), is not curative therapy. New approaches to prevent relapse after AHCT and to treat relapse are needed.
* In murine models, we used ex vivo culture to generate rapamycin-resistant, Th1 (type 1 T helper cells)/Tc1 (T cytotoxic cells, type 1) polarized T cells (Th1/Tc1.Rapamycin (Rapa) cells) that were both rapamycin-resistant and apoptosis-resistant with an increased in vivo survival and in vivo function.
* Because Th1 /Tc1 polarized lymphocytes are pivotal in anti-tumor effects, we hypothesize that adoptive transfer of Th1/Tc1Rapa cells will be of benefit to MM patients.

Objectives:

Primary

Dose escalation study

Evaluate the feasibility and toxicity of an infusion of autologous, ex vivo rapamycin-generated, anti-cluster of differentiation 3 (CD3) and anti-cluster of differentiation 28 (CD28) co-stimulated, Th1/Tc1 lymphocytes (Th1/Tc1.Rapa cells) in subjects diagnosed with high-risk multiple myeloma following AHCT.

MM Relapse Prevention and Treatment Cohorts

* For Cohort A, in newly diagnosed MM patients who have received AHCT, evaluate the safety of a defined regimen of Th1/Tc1.Rapa cell therapy and determine progression-free survival.
* For Cohort B, in relapsed MM, determine the partial response (PR)/complete response (CR) rate of Th1/Tc1.Rapa cell therapy.

Eligibility:

* For Cohort A relapse prevention, patients with MM (normal- or high-risk) who are receiving induction therapy and subsequent AHCT.
* For Cohort B relapse therapy, patients with MM who have measurable disease after at least 2 prior treatment regimens.

Design:

* For Cohort A, patients will receive two infusions of autologous Th1/Tc1.Rapa cells (at one and two months post-AHCT; each infusion preceded by a 7-day course of immune modulating chemotherapy [pentostatin plus low-dose cyclophosphamide; PC regimen].
* For Cohort B relapse therapy, patients will up to four infusions of Th1/Tc1.Rapa cells, with each infusion preceded by either a 7-day or 14-day PC regimen.

ELIGIBILITY:
* INCLUSION CRITERIA:

MULTIPLE MYELOMA CRITERIA:

Criteria for Cohort A (recently diagnosed subjects; to receive autologous hematopoietic cell transplantation (AHCT)):

* Must have presence of clonal plasma cells in the bone marrow greater or equal to 10% or biopsy proven plasmacytoma
* Must have either:

  1. presence of an M-component (Immunoglobulin G (IgG) or Immunoglobulin G (IgA)) in serum greater or equal to 1g/dl or in urine greater or equal to 200 mg/24 h; or
  2. presence of an abnormal serum free light chain (FLC) ratio on the serum FLC assay.

Criteria for Cohort B (multiply relapsed multiple myeloma):

* Must have measurable multiple myeloma (MM), as defined by: serum M-protein greater than or equal to 1 g/dL, urine M-protein greater than or equal to 200 mg/24 hours, involved serum free light chain (FLC) level greater than or equal to 10 mg/dL, biopsy proven plasmacytoma, or more than 30% bone marrow plasma cells.
* Must have received at least 2 different treatment regimens for MM.

Other eligibility criteria (applies to both Cohort A and Cohort B, unless specified):

* Age greater than or equal to 18 years and less than or equal to 75 years. In subjects between 65 and 75 years of age, physiologic age and co-morbidity will be thoroughly evaluated before enrolling. Specifically, any history of cardio-vascular pathology or symptoms, not clearly fitting the exclusion criteria will prompt an evaluation by a Clinical Center Cardiologist and eligibility will be considered on a case-by-case basis.
* For Cohort A only, high-dose chemotherapy and AHCT must be planned; with amendment K, post-transplant maintenance therapy will not be permitted.
* Karnofsky performance status (KPS) of 70% or greater. Lower KPS down to 50% may be acceptable if the restriction of activity is solely due to intractable pain from myeloma lesions.
* Ejection fraction (EF) by multi-gated acquisition scan (MUGA) or two-dimensional (2-D) echocardiogram within institution normal limits. In case of low EF, the subject may remain eligible after a stress echocardiogram is performed if the EF is more than 35% and if the increase in EF with stress is estimated at 10% or more.
* Serum creatinine less than or equal to 2.5 mg/dl,
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 times the upper limit of normal.
* Bilirubin less than or equal to1.5 (except if due to Gilbert's disease).
* Corrected carbon monoxide diffusing capacity (DLCO) greater than or equal to 50% on Pulmonary Function Tests
* No history of abnormal bleeding tendency or predisposition to repeated infections.
* Patients must be able to give informed consent

EXCLUSION CRITERIA:

* Prior allogeneic stem cell transplantation
* Hypertension not adequately controlled by 3 or less medications.
* History of cerebro-vascular accident within 6 months of enrollment.
* History of documented pulmonary embolus within 6 months of enrollment.
* Clinically significant cardiac pathology: myocardial infarction within 6 months prior to enrollment, Class III or IV heart failure according to New York Heart Association (NYHA), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patients with a history of coronary artery bypass grafting or angioplasty will receive a cardiology evaluation and be considered on a case-by-case basis.
* Human immunodeficiency virus (HIV) seropositive
* Patients known or found to be pregnant or who is unwilling to stop breast-feeding.
* Patients of childbearing age who are unwilling to practice contraception or other means of avoiding pregnancy.

Patients may be excluded at the discretion of the principal investigator (PI) if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-11-10 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health (NIH) Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Background] Tosi P, Zamagni E, Cellini C, Plasmati R, Cangini D, Tacchetti P, Perrone G, Pastorelli F, Tura S, Baccarani M, Cavo M. Neurological toxicity of long-term (>1 yr) thalidomide therapy in patients with multiple myeloma. Eur J Haematol. 2005 Mar;74(3):212-6. doi: 10.1111/j.1600-0609.2004.00382.x. PMID 15693790
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0016.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the planned protocol cohort 7, no patients were accrued due to lack of feasibility in terms of T cell manufacturing. That is, cohort 6 evaluated 15X10EE6 cells per kg, which was the max. number that could be manufactured due to limiting reagents for cell culture. 3/34 pts signed consent but did not receive therapy due to progressive malignancy.
Groups:
- Cohort 1 - 1x10(5) T Cells/kg: 1x10(5) Th1/Tc1 Rapa cells/kg of body weight
- Cohort 2 - 5x10(5) T Cells/kg: 5x10(5) Th1/Tc1 Rapa cells/kg of body weight
- Cohort 3 - 1x10(6) T Cells/kg: 1x10(6) Th1/Tc1 Rapa cells/kg of body weight
- Cohort 4 - 3x10(6) T Cells/kg: 3x10(6) Th1/Tc1 Rapa cells/kg of body weight
- Cohort 5 - 5x10(6) T Cells/kg: 5x10(6) Th1/Tc1 Rapa cells/kg of body weight
- Cohort 5B - 5x10(6) T Rapa Cells/kg: 5x10(6) Th1/Tc1 Rapa cells/kg of body weight; Three sequential infusions with at least two months between infusions.
- Cohort 6 - 15x10(6) T Cells/kg: 15x10(6) Th1/Tc1 Rapa cells/kg of body weight
- Cohort 7 - 45x10(6) T Cells/kg of: 45x10(6) Th1/Tc1 Rapa cells/kg of body weight
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1/Tc1 Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1 Rapa Cells: Six Th1.rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1Rapa: 5 x 10e(6) cells/kg
- Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma: Th1/Tc1.Rapa for Relapsed Multiple Myeloma
  Adoptive Immunotherapy: Th1/Tc1 Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1rapa: 5 x 10e(6) cells/kg
Period: Overall Study
Arm/Group | Cohort 1 - 1x10(5) T Cells/kg | Cohort 2 - 5x10(5) T Cells/kg | Cohort 3 - 1x10(6) T Cells/kg | Cohort 4 - 3x10(6) T Cells/kg | Cohort 5 - 5x10(6) T Cells/kg | Cohort 5B - 5x10(6) T Rapa Cells/kg | Cohort 6 - 15x10(6) T Cells/kg | Cohort 7 - 45x10(6) T Cells/kg of | Cohort A - Th1/Tc1.Rapa Prevention of Relapse | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma
Started | 2 | 1 | 1 | 2 | 7 | 5 | 7 | 0 | 1 | 5
Completed | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1
Not Completed | 2 | 1 | 1 | 1 | 5 | 4 | 6 | 0 | 0 | 4
Not completed — Principal investigator discretion | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Not completed — Disease progression on study | 1 | 1 | 1 | 1 | 4 | 2 | 5 | 0 | 0 | 2
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the planned protocol cohort 7, no patients were accrued due to lack of feasibility in terms of T cell manufacturing. That is, cohort 6 evaluated 15X10EE6 cells per kg, which was the maximum number that could be manufactured due to limiting reagents for cell culture.
Groups:
- Cohort 1 - 1x10(5) T Cells/kg: 1x10(5) Th1/Tc1.Rapa cells/kg of body weight
- Cohort 2 - 5x10(5) T Cells/kg: 5x10(5) Th1/Tc1.Rapa cells/kg of body weight
- Cohort 3 - 1x10(6) T Cells/kg: 1x10(6) Th1/Tc1.Rapa cells/kg of body weight
- Cohort 4 - 3x10(6) T Cells/kg: 3x10(6) Th1/Tc1.Rapa cells/kg of body weight
- Cohort 5 - 5x10(6) T Cells/kg: 5x10(6) Th1/Tc1.Rapa cells/kg of body weight
- Cohort 5B - 5x10(6) T Rapa Cells/kg: 5x10(6) Th1/Tc1.Rapa cells/kg of body weight; Three sequential infusions with at least two months between infusions.
- Cohort 6 - 15x10(6) T Cells/kg: 15x10(6) Th1/Tc1.Rapa cells/kg of body weight
- Cohort 7 - 45x10(6) T Cells/kg: 45x10(6) Th1/Tc1.Rapa cells/kg of body weight
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1/Tc1.Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1 Cells: Six Th1/Tc1.Rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/TC1 Rapa Cell Therapy: Th1/TC1rapa: 5 x 10e(6) cells/kg
- Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma: Th1/Tc1.Rapa for Relapsed Multiple Myeloma
  Adoptive Immunotherapy: Th1/Tc1.Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Th1/TC1 Rapa Cell Therapy: Th1/Tc1.Rapa: 5 x 10e(6) cells/kg
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 1x10(5) T Cells/kg | Cohort 2 - 5x10(5) T Cells/kg | Cohort 3 - 1x10(6) T Cells/kg | Cohort 4 - 3x10(6) T Cells/kg | Cohort 5 - 5x10(6) T Cells/kg | Cohort 5B - 5x10(6) T Rapa Cells/kg | Cohort 6 - 15x10(6) T Cells/kg | Cohort 7 - 45x10(6) T Cells/kg | Cohort A - Th1/Tc1.Rapa Prevention of Relapse | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma | Total
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 7 | 5 | 7 | 0 | 1 | 5 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 0 | 2 | 4 | 5 | 4 | 0 | 0 | 2 | 20
  >=65 years | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 0 | 1 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.58) | 41.3 (0) | 65.8 (0) | 46.7 (15.56) | 58.19 (13.79) | 57.64 (6.18) | 59.29 (9.58) |  | 66.9 (0) | 63.6 (9.08) | 55.8 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 2 | 4 | 3 |  | 1 | 4 | 18
  Male | 1 | 0 | 0 | 1 | 5 | 1 | 4 |  | 0 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 2 | 1 | 1 | 2 | 7 | 5 | 6 |  | 1 | 4 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 2 | 1 | 0 |  | 0 | 1 | 5
  White | 1 | 0 | 1 | 1 | 5 | 4 | 5 |  | 1 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 2 |  | 0 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 1 | 2 | 7 | 5 | 7 |  | 1 | 5 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Adverse Event Attributable to the Investigational Therapy
Description: Participants were assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Time Frame: 2 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5B - - 5x10(6) T Cells/kg: 5x10(6) Th1/Tc1.Rapa cells/kg of body weight; Three sequential infusions with at least two months between infusions.
- Cohort 6 - 15x10(6) T Cells/kg: 15x10(6) Th1/Tc1.Rapac ells/kg of body weight
- Cohort 7- 45x10(6) T Cells/kg: 45x10(6) Th1/Tc1.Rapa cells/kg of body weight
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1/Tc1.Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1 Cells: Six Th1/Tc1.Rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1.Rapa 5 x 10e(6) cells/kg
- Cohort B - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa for Relapsed Multiple Myeloma
  Adoptive Immunotherapy: Th1.rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1.Rapa: 5 x 10e(6) cells/kg
Arm/Group | Cohort 1 - 1x10(5) T Cells/kg | Cohort 2 - 5x10(5) T Cells/kg | Cohort 3 - 1x10(6) T Cells/kg | Cohort 4 - 3x10(6) T Cells/kg | Cohort 5 - 5x10(6) T Cells/kg | Cohort 5B - - 5x10(6) T Cells/kg | Cohort 6 - 15x10(6) T Cells/kg | Cohort 7- 45x10(6) T Cells/kg | Cohort A - Th1/Tc1.Rapa Prevention of Relapse | Cohort B - Th1/Tc1.Rapa Prevention of Relapse
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 7 | 5 | 7 | 0 | 1 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Progression Free Survival in Cohort A Th1 (Type 1 T Helper Cells)/Tc1 (T Cytotoxic Cells, Type 1) Rapa Prevention of Relapse
Description: Progressive disease is assessed by the Consensus of the International Myeloma Working Group criteria and is defined as one or more of the following: Increases of greater or equal to 25% in serum M-component (minimum absolute increase of 0.5 g/dl) or urine M-component (minimum absolute increase of 200mg/24h) or percentage of bone marrow plasma cells (minimum absolute percentage of 10%) or size of bone lesions or new plasmacytoma, or development of hypercalcemia solely attributable to the disease.
Time Frame: Study completion at 22 months
Population: The PFS was only used in cohort A, which had just one patient.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1 (type 1 T helper cells)/Tc1 (T cytotoxic cells, type 1) Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1.Rapa Cells: Six Th1.rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1.Rapa: 5 x 10e(6) cells/kg
Arm/Group | Cohort A - Th1/Tc1.Rapa Prevention of Relapse
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: Number of Patients Who Developed a Partial Response (PR)+Complete Response (CR) in Cohort B at Any Time Point Post Therapy With PR/CR Being Maintained Until Study Completed
Description: Patients whose tumors shrunk and were disease free after therapy in cohort B. Partial response and complete response were assessed by the Consensus of the International Myeloma Working Group criteria. Partial response is defined as 50% or greater reduction in serum M-protein and 90% or greater reduction in 24-h urinary M-protein (or to less than 200 mg per 24h), 50% or greater reduction in the size of soft tissue plasmacytomas, if present at baseline, no evidence of progressive or new bone lesions if radiographic studies were performed (X-rays not required in absence of clinical indication). Complete response is defined as negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and 5% or less plasma cells in bone marrow and no evidence of progressive or new bone lesion if radiographic studies were performed. Progressive disease is increases of ≥25% in serum M-component/urine M-component, or size of bone lesions.
Time Frame: Study completion at 22 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma: Th1/Tc1.Rapa for Relapsed Multiple Myeloma
  Adoptive Immunotherapy: Th1 (type 1 T helper cells)/Tc1 (T cytotoxic cells, type 1) Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1.Rapa: 5 x 10e(6) cells/kg
Arm/Group | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma
Number analyzed (Participants) | 5
Participants | 2

4. Secondary Outcome: Immune Reconstitution in Recipients of Th1.(T Helper Cell) Rapa Cells.
Description: Immune reconstitution in recipients of Th1.rapa cells was determined by flow cytometry.
Time Frame: Baseline, prior to chemotherapy, and 2 weeks, 1, 2, and 3 months after final T cell infusion
Population: For the planned protocol cohort 7, no pts were accrued due to lack of feasibility in terms of T cell manufacturing. That is, cohort 6 evaluated 15X10EE6 cells per kg, which was the max. # that could be manufactured due to limiting reagents for cell culture. Outcome measure not done; data not collected in real-time due to premature closure of study.
Groups:
- Cohort 5B - 5x10(6) Th1 Rapa Cells/kg: 5x10(6) Th1 rapa cells/kg of body weight; Three sequential infusions with at least two months between infusions.
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1/Tc1.Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1 Cells: Six Th1/Tc1.Rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/Tc1 Rapa Cell Therapy: Th1/Tc1.Rapa: 5 x 10e(6) cells/kg
Arm/Group | Cohort 1 - 1x10(5) T Cells/kg | Cohort 2 - 5x10(5) T Cells/kg | Cohort 3 - 1x10(6) T Cells/kg | Cohort 4 - 3x10(6) T Cells/kg | Cohort 5 - 5x10(6) T Cells/kg | Cohort 5B - 5x10(6) Th1 Rapa Cells/kg | Cohort 6 - 15x10(6) T Cells/kg | Cohort 7 - 45x10(6) T Cells/kg | Cohort A - Th1/Tc1.Rapa Prevention of Relapse | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to last date off study, 81 months and 6 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 5B - 5x10(6) T Cells/kg: 5x10(6) Th1/Tc1.Rapa cells/kg of body weight; Three sequential infusions with at least two months between infusions.
- Cohort 7 - 45x10(6) T Cells/kg: 45x10(6) th1 cells/kg of body weight
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1.rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1 Cells: Six Th1.rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/TC1 Rapa Cell Therapy: Th1/TC1rapa: 5 x 10e(6) cells/kg
- Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma: Th1/Tc1.Rapa for Relapsed Multiple Myeloma
  Adoptive Immunotherapy: Th1.rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Th1/TC1 Rapa Cell Therapy: Th1/TC1rapa: 5 x 10e(6) cells/kg
Arm/Group | Cohort 1 - 1x10(5) T Cells/kg | Cohort 2 - 5x10(5) T Cells/kg | Cohort 3 - 1x10(6) T Cells/kg | Cohort 4 - 3x10(6) T Cells/kg | Cohort 5 - 5x10(6) T Cells/kg | Cohort 5B - 5x10(6) T Cells/kg | Cohort 6 - 15x10(6) T Cells/kg | Cohort 7 - 45x10(6) T Cells/kg | Cohort A - Th1/Tc1.Rapa Prevention of Relapse | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma
Number analyzed (Participants) | 2 | 1 | 1 | 2 | 7 | 5 | 7 | 0 | 1 | 5
Participants | 1 | 1 | 1 | 2 | 5 | 2 | 3 | 0 | 1 | 4

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to last date off study, 81 months and 6 days.
Description: For the planned protocol cohort 7, no patients were accrued due to lack of feasibility in terms of T cell manufacturing. That is, cohort 6 evaluated 15X10EE6 cells per kg, which was the maximum number that could be manufactured due to limiting reagents for cell culture.
Groups:
- Cohort A - Th1/Tc1.Rapa Prevention of Relapse: Th1/Tc1.Rapa Prevention of Relapse
  Adoptive Immunotherapy: Th1/Tc1.Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Rapamycin-Generated Autologous Th1/Tc1 Cells: Six Th1.rapa cell doses will be tested in cohorts of 1-6 subjects each: ranging from 10e(5) to 15 x 10e(6) cells/kg of body weight.
  Th1/TC1 Rapa Cell Therapy: Th1/TC1rapa: 5 x 10e(6) cells/kg
- Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma: Th1/Tc1.Rapa for Relapsed Multiple Myeloma
  Adoptive Immunotherapy: Th1/Tc1.Rapa cell infusion will be evaluated after administration of a 7-day or 14-day course of immune depleting chemotherapy (pentostatin plus cyclophosphamide regimen).
  Th1/TC1 Rapa Cell Therapy: Th1/TC1rapa: 5 x 10e(6) cells/kg
Arm/Group | Cohort 1 - 1x10(5) T Cells/kg | Cohort 2 - 5x10(5) T Cells/kg | Cohort 3 - 1x10(6) T Cells/kg | Cohort 4 - 3x10(6) T Cells/kg | Cohort 5 - 5x10(6) T Cells/kg | Cohort 5B - 5x10(6) T Rapa Cells/kg | Cohort 6 - 15x10(6) T Cells/kg | Cohort 7 - 45x10(6) T Cells/kg | Cohort A - Th1/Tc1.Rapa Prevention of Relapse | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/2 | 0/7 | 0/5 | 1/7 | 0/0 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/1 | 0/2 | 1/7 | 0/5 | 1/7 | 0/0 | 0/1 | 1/5
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 1/1 | 2/2 | 5/7 | 2/5 | 3/7 | 0/0 | 1/1 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 1x10(5) T Cells/kg (N=2) | Cohort 2 - 5x10(5) T Cells/kg (N=1) | Cohort 3 - 1x10(6) T Cells/kg (N=1) | Cohort 4 - 3x10(6) T Cells/kg (N=2) | Cohort 5 - 5x10(6) T Cells/kg (N=7) | Cohort 5B - 5x10(6) T Rapa Cells/kg (N=5) | Cohort 6 - 15x10(6) T Cells/kg (N=7) | Cohort 7 - 45x10(6) T Cells/kg (N=0) | Cohort A - Th1/Tc1.Rapa Prevention of Relapse (N=1) | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma (N=5)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 1x10(5) T Cells/kg (N=2) | Cohort 2 - 5x10(5) T Cells/kg (N=1) | Cohort 3 - 1x10(6) T Cells/kg (N=1) | Cohort 4 - 3x10(6) T Cells/kg (N=2) | Cohort 5 - 5x10(6) T Cells/kg (N=7) | Cohort 5B - 5x10(6) T Rapa Cells/kg (N=5) | Cohort 6 - 15x10(6) T Cells/kg (N=7) | Cohort 7 - 45x10(6) T Cells/kg (N=0) | Cohort A - Th1/Tc1.Rapa Prevention of Relapse (N=1) | Cohort B - Th1/Tc1.Rapa for Relapsed Multiple Myeloma (N=5)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (4) | 1 (7) | 1 (3) | 1 (3) | 2 (10) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (9) | 1 (6) | 1 (2) | 0 (0) | 4 (7) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CPK increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
3/34 pts signed consent but never received therapy due to progressive malignancy that precluded their ability to receive the experimental therapy. These participants were not assigned to a cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT01239368/Prot_SAP_000.pdf
  • Informed Consent Form (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT01239368/ICF_001.pdf